CLINICAL TRIAL: NCT03859245
Title: Photobiomodulation & Ketogenic Diet for Treatment of Mid-periphery Retinal Disorders (Diabetic Retinopathy, Dry AMD, Hard Drusen Formation) for Alzheimer's Disease Prevention
Brief Title: Photobiomodulation & Ketogenic Diet for Treatment of Mid-periphery Retinal Disorders for Alzheimer's Disease Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bristlecone Health, Inc. (Industry)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bristlecone-002
Record Dates: First submitted 2019-02-24; First posted 2019-03-01 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Diabetic Retinopathy (DR); Age-related Macular Degeneration (AMD); Mid-peripheral Drusen Formation; Diabetic Macular Edema (DME)
Keywords: Photobiomodulation; Diabetic Retinopathy (DR); Age-related Macular Degeneration (AMD); Mid-peripheral Drusen; Alzheimer's disease (AD); Ketogenic Diet (KD)
MeSH Terms: conditions — Diabetic Retinopathy; Macular Degeneration; Alzheimer Disease | interventions — Low-Level Light Therapy; Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: To assess differences between the control and experimental groups, a mixed model will be fit for each variable separately using both baseline (week 0) and post program (week 36) values for each subject. Models will include week, group, and their interaction as fixed effects, gender as a covariate, and subject as random effect. To assess significant differences, we will use the difference at week 36 adjusted for the baseline difference, report p-values, least squares mean, and 95% confidence intervals. Further analysis of treatment effects over time will be examined by comparing the within-group differences over time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Subjects in the experimental group will receive clinically prescribed meal plans designed to facilitate prolonged benign dietary ketosis (BDK) purposed at glucose regulation, improved insulin sensitivity and restored metabolic flexibility. Photobiomodulation therapy, via Joovv red light/infrared LED device, will be administered three times per week, 20 minutes per session.
  Interventions: Behavioral: Photobiomodulation; Behavioral: Ketogenic diet
- Control group (Active Comparator): Subjects in the control group will follow current dietary protocol (Standard American Diet- SAD). Photobiomodulation therapy,via Joovv red light/infrared LED device, will be administered three times per week, 20 minutes per session.
  Interventions: Behavioral: Photobiomodulation

INTERVENTIONS:
Behavioral: Photobiomodulation — Photobiomodulation therapy, via Joovv red light/infrared LED device, three days/week, 20 minutes per session for experimental and control groups.
Behavioral: Ketogenic diet — Experimental group will follow a clinically prescribed ketogenic diet.
  Arms: Experimental group

SUMMARY:
The study will explore the impact of photobiomodulation (PBM), pulsating at frequencies of red (660nm) and near-infrared (810nm)(NIR), concurrent with a ketogenic dietary protocol (serum ketones @ .5 - 2.0 mmol/L) to mediate vascular features of diabetic retinopathy (DR), diabetic macular edema (DME), age-related macular degeneration (AMD), mid-peripheral drusens, visual acuity and retinal disorders. Red and near-infrared light via light-emitting diode (LED) treatment promotes retinal healing and improves visual acuity by augmenting cellular energy metabolism, enhancing mitochondrial function, increasing cytochrome C oxidase activity, stimulating antioxidant protective pathways and promoting cell survival. LED therapy directly benefits neurons in the retina, the lateral geniculate nucleus and the visual cortex; likewise, a ketogenic dietary protocol shows metabolic and neuro-modulatory benefits within the CNS, most notably as treatment for refractory epilepsy. Photobiomodulation has been approved as a non-significant risk (NSR) modality for the treatment of eye disorders.

DETAILED DESCRIPTION:
As part of the central nervous system (CNS), the retina shares key structural and functional features with the brain, making it a potential portal into a patient's medical future. Since the cerebral and retinal microvasculature are strikingly similar, the condition of retinal vasculature has been considered a proxy for cerebral vascular health. Retinal nerve fiber layer thinning, loss of retinal ganglion cells and optic disc changes may be associated with Alzheimer's disease (AD). Additionally, drusen formation in the macula has been shown to potentially predict AD severity. While the macula has been the primary focus of research for retinal abnormalities, the peripheral retina may be the earliest predictor of neurodegeneration via dry AMD (age-related macular degeneration) and diabetic retinopathy (DR). Ultra-widefield (UWF) retinal imaging has been shown to identify early biomarkers for AD and its progression. Peripheral hard drusen formation and changes to the vasculature beyond the posterior pole are associated with the pathogenesis of AD. A recent clinical trial found a significantly higher prevalence of the hard drusen phenotype within the periphery of AD patients (14/55; 25.4%) compared to controls (2/48; 4.2%)[p = 0.04]. Analyzing the peripheral retina for biomarkers of neurodegeneration such as drusen formation and vascular pathology offers a foundational diagnostic standard for preventative care. The proposed intervention purposes to inhibit the pro-inflammatory cascade in the retinal and cerebral vasculature via restoration of mitochondrial signaling, metabolic substrate flexibility and reduction of oxidative stress using a clinically prescribed ketogenic dietary protocol concurrent with photobiomodulation.

Deterioration in metabolic energy pathways is a prominent feature of AD, Parkinson's disease (PD), retinitis pigmentosa (RP), diabetic retinopathy, dry AMD, glaucoma and cerebellar atrophy. Common etiological mechanisms of neurodegenerative disorders of the eye and the CNS include mutations in the DJ-1 and Myc-Modulator (MM-1) genes and impaired mitochondrial signaling. Photobiomodulation (PBM) therapy, pulsating frequencies of 660nm and 810nm, has been shown to generate vasoprotective, neuroprotective, immunomodulatory and regenerative effects on mitochondrial function, cellular respiration, and improve retinal and cerebral vascularity. Recent studies have shown significant outcomes using PBM in the treatment of AMD, diabetic retinopathy, Stargardt disease, Leber's hereditary optic neuropathy, Parkinson's disease and Alzheimer's disease. Common to the etiology of each of these disease states is oxidative stress, an inflammatory cascade and activation of apoptotic pathways. Photobiomodulation proves to be both pro-oxidant in the short-term and antioxidant in the long term to potentiate a hormetic dose response. Likewise, PBM modulates inflammation via the immune regulatory pathways, reduces risk for retinal vascular dysfunction and offers protection from photoreceptor cell death. In primary astrocytes, improved immune regulation attenuates cerebral inflammation and oxidative stress induced by beta amyloid and initiates reparative action on protein misfolding by activating/modulating metabolic control over folding/unfolding.

Neuro-modulatory outcomes are well documented for ketogenic nutritional protocols; most recently, dietary ketosis has been shown to mediate Type 2 Diabetes Mellitus (T2DM), significantly reduce systemic inflammation, restore endocrine homeostasis and improve peripheral and cerebral insulin sensitivity. A recent study demonstrating the neuroprotective effects of a ketogenic diet on glaucoma suggests that increased insulin sensitivity protects retinal ganglion cell structure and function, reduces NF-KB p65 nuclear translocation and inhibits expression of pro-inflammatory molecules. The 8-week ketogenic nutritional intervention resolved energy demand and ameliorated inflammation by stimulating HCAR1-ARRB2 (Hydroxycarboxylic acid receptors-Arrestin beta -2) signaling pathways.

The rapidly increasing demand for healthcare among America's aging population warrants novel, integrative strategies focused on non-invasive treatments to ensure patient compliance and maximize health span concurrent with lifespan. Photobiomodulation therapy combined with multidisciplinary lifestyle modifications, such as ketogenic nutritional protocols, offered to patients in the optometry setting provides a viable therapeutic approach for healthcare providers on the front-line of diabetes care. The PBM intervention features both a diagnostic tool for prevention and a treatment model for retinal/cerebral microvasculature diseases common to aging: AD, PD, diabetic retinopathy, AMD, glaucoma and retinitis.

The study will explore the impact of photobiomodulation, pulsating at frequencies of red (660nm) and near-infrared (810nm), concurrent with a ketogenic dietary protocol (serum ketones @ .5 - 2.0 mmol/L) to mediate vascular features of diabetic retinopathy, diabetic macular edema, age-related macular degeneration (AMD), mid-peripheral drusens, visual acuity and retinal disorders. Red and near-infrared light (NIR) via light-emitting diode (LED) treatment promotes retinal healing and improves visual acuity by augmenting cellular energy metabolism, enhancing mitochondrial function, increasing cytochrome C oxidase activity, stimulating antioxidant protective pathways and promoting cell survival. LED therapy directly benefits neurons in the retina, the lateral geniculate nucleus and the visual cortex; likewise, a ketogenic dietary protocol shows metabolic and neuro-modulatory benefits within the CNS, most notably as treatment for refractory epilepsy. Photobiomodulation has been approved as a non-significant risk (NSR) modality for the treatment of eye disorders.

ELIGIBILITY:
Inclusion Criteria:

Male or Female (age 18-80)

Previously diagnosed with MetS and/or T2DM as measured by possessing at least 2 of the following physiological measures: type II diabetes, BMI >30, HgA1c > 5.7, waist/height ratio >.6, fasting glucose > 125

Previously diagnosed with at least one of the following: mid-peripheral drusen formation, diabetic retinopathy (DR), age-related macular degeneration (AMD) or diabetic macular edema

Exclusion Criteria:

Previously diagnosed with Alzheimer's disease (AD), dementia or Parkinson's disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02-23 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Diabetic Retinopathy (DR) pathology | 36 weeks
  Improvement in number and severity of hemorrhages and hard and soft exudates as measured by the Daytona Plus (Panoramic Ophthalmoscope P200T)
Diabetic Macular Edema (DME) pathology | 36 weeks
  Lower incidence of macular edema as measured by Optos Daytona Plus (Panoramic Ophthalmoscope P200T) and Optovue XR Avanti 3 OCT (Ocular Coherence Tomography) Imaging Systems
Dry Age-related Macular Degeneration (AMD) pathology | 36 weeks
  Reduction in size and number of drusen in early and intermediate stages of Dry AMD pathology as measured byOptos Daytona Plus (Panoramic Ophthalmoscope P200T) and Optovue XR Avanti 3 OCT (Ocular Coherence Tomography) Imaging Systems
Hard Drusen in the Mid-periphery pathology | 36 weeks
  Reduction in size and/or density of drusen as measured by the Optos Daytona Plus (Panoramic Ophthalmoscope P200T)

SECONDARY OUTCOMES:
HgA1c | 36 weeks
  Assessment of changes in HgA1c (Hemoglobin A1c) over time. Ranges: <5.7%
Fasting Insulin | 36 weeks
  Assessment of changes in fasting insulin over time. Ranges: < 2.6-11.1 mU/L
Fasting Glucose | 36 weeks
  Assessment of changes in fasting glucose over time. Ranges 74-100 mg/dL
HOMA-IR | 36 weeks
  Assessment of changes in HOMA-IR over time. Ranges <1.0
Triglycerides/HDL ratio | 36 weeks
  Assessment of changes in triglycerides/HDL ratio over time. Ranges <2.0

CONTACTS AND LOCATIONS:
Locations (1):
- Yankee Eye Clinic, Eagan, Minnesota, United States